CLINICAL TRIAL: NCT04200404
Title: A Phase Ib/II, Multicenter Open-label Study of CS1001 in Combination With Regorafenib in Patients With Advanced or Refractory Solid Tumors
Brief Title: A Study of CS1001 in Combination With Regorafenib in Patients With Advanced or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CStone Pharmaceuticals (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS1001/Regorafenib-101
Record Dates: First submitted 2019-12-13; First posted 2019-12-16 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Advanced Refractory Solid Tumors
MeSH Terms: interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase Ib arm (Experimental): arms 1. Phase Ib: advanced or refractory solid tumors;
  Interventions: Drug: CS1001; Drug: Regorafenib
- Phase II arm (Experimental): arms 2.Phase II: subjects with tumor of specific types
  Interventions: Drug: CS1001; Drug: Regorafenib

INTERVENTIONS:
Drug: CS1001 — One course will last 28 days. CS1001 will be intravenously administered every 4 weeks (Q4W).
Drug: Regorafenib — One course will last 28 days. Administration will be orally (p.o.) taken at different dose schemes.
  Other Names: BAY 73-4506

SUMMARY:
This is a multicenter, open-label study of CS1001 in combination with regorafenib in participants with advanced or refractory cancers. There will be a dose escalation portion in "allcomers"to find a suitable dose of regorafenib for combination use with CS1001. This study will also enroll participants with specific tumor types in the phase II part of the study to assess the efficacy, pharmacokinetics and safety of the combined regimen (RP2D of regorafenib + CS 1001)

ELIGIBILITY:
Inclusion Criteria:

* All participants must have unresectable advanced or metastatic tumors that have histologic or cytologic documentation confirmed.
* Participant must have at least one measurable lesion by CT or MRI per RECIST 1.1; radiographic tumor assessment should be performed within 28 days prior to initiation of study treatment.
* ECOG performance status score of 0 or 1.
* Life expectancy ≥ 12 weeks.
* Fresh or archival tumor tissue must be provided for PD-L1 expression testing in selected cohorts.
* Adequate organ function
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test result. Either Female or male participants must agree to use adequate contraceptive measures from signing informed consent and for 180 days after last investigational product administration, except for a participant with documented surgical sterilization or a postmenopausal female.
* Any toxic effects of prior anti-cancer therapy or surgical procedures resolved to baseline severity or NCI-CTCAE version 5 Grade 1 (except alopecia or other toxicities not considered a safety risk for the patient at investigator's discretion).
* Subjects with hepatitis B virus (HBV) infection must have HBV DNA < 2000 IU/mL at screening, and requires continue anti-HBV treatment in the study

Exclusion Criteria:

* Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured.
* Participants with any condition that impairs their ability to take oral medication, such as lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome.
* Has known central nervous system (CNS) metastases and/or carcinomatous meningitis that is either symptomatic or untreated.
* Any prior (within 1 year) or current clinically significant ascites as measured by physical examination and that requires active paracentesis for control.
* Significant history of cardiac disease within 6 months prior to Day 1 of Cycle 1, myocardial infarction within the previous year, or current cardiac ventricular arrhythmias requiring medication, or left ventricular ejection fraction (LVEF) is below 50%.
* History or evidence of poorly controlled arterial hypertension.
* Any serious or uncontrolled medical disorder or active infection may increase the risk associated with study participation or dose.
* Administration of drugs known as strong CYP3A4 inducers or strong CYP3A4 inhibitors and the last dose was given in < 5 half-lives from the first investigational product administration.
* Any hemorrhage or bleeding event ≥ CTCAE Grade 3 within 28 days prior to the start of study treatment.

Other inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2021-05-13 (Actual); Study Completion 2021-08-18 (Actual)

PRIMARY OUTCOMES:
Phase Ib (Safety Evaluation): Number of participants with adverse events | Baseline up to 90 days post last dose, up to 2 years
Phase Ib (Safety Evaluation): Dose Limiting Toxicity (DLT) | Baseline up to 90 days post last dose, up to 2 years
Phase II (Efficacy Expansion): Objective response rate (ORR) | Up to 2 years

SECONDARY OUTCOMES:
Phase Ib (Safety Evaluation): Objective response rate (ORR) | Up to 2 years
Phase Ib (Safety Evaluation) and/or Phase II (Efficacy Expansion): Disease control rate (DCR) | Up to 2 years
Phase Ib (Safety Evaluation) and/or Phase II (Efficacy Expansion): Progression Free Survival (PFS) | Up to 2 years
Phase Ib (Safety Evaluation) and/or Phase II (Efficacy Expansion): Duration of Response (DoR) | Up to 2 years
Phase Ib (Safety Evaluation) and/or Phase II (Efficacy Expansion): Overall Survival (OS) | Up to 2 years
Phase Ib (Safety Evaluation) and/or Phase II (Efficacy Expansion): Occurrence of anti-CS1001 antibody | From first dose to 30 days after last dose, up to 2 years
Phase II (Efficacy Expansion): : Number of participants with adverse events | Baseline up to 90 days post last dose, up to 2 years
Phase Ib (Safety Evaluation) and/or Phase II (Efficacy Expansion): Area under the plasma concentration-time curve (AUC)0-t of CS1001 | From first dose to 30 days after last dose, up to 2 years
Phase Ib (Safety Evaluation) and/or Phase II (Efficacy Expansion): Maximum plasma concentration (Cmax) of CS1001 | From first dose to 30 days after last dose, up to 2 years
Phase Ib (Safety Evaluation) and/or Phase II (Efficacy Expansion): Time to reach maximum plasma concentration (Tmax) of CS1001 | From first dose to 30 days after last dose, up to 2 years
Phase Ib (Safety Evaluation) and/or Phase II (Efficacy Expansion): Terminal elimination half-life (t1/2) of CS1001 | From first dose to 30 days after last dose, up to 2 years
Phase Ib (Safety Evaluation) and/or Phase II (Efficacy Expansion): Clearance at Steady State (CLss) of CS1001 | From first dose to 30 days after last dose, up to 2 years
Phase Ib (Safety Evaluation): Maximum plasma concentration (Cmax) of regorafenib | From first dose to 30 days after last dose, up to 2 years
Phase Ib (Safety Evaluation): Minimum plasma concentration (Cmin) of regorafenib | From first dose to 30 days after last dose, up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Ashford Cancer Centre Research, Kurralta Park, South Australia, Australia